CLINICAL TRIAL: NCT05036486
Title: The Registry of Genetic Alterations of Taiwan Biliary Tract Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Tri-Service General Hospital (Other); Chang Gung Medical Foundation (Linkou Branch) (Unknown); Taipei Medical University Shuang Ho Hospital (Other); Koo Foundation Sun Yat-Sen Cancer Center (Other); China Medical University Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Medical University Chung-Ho Memorial Hospital (Other); Chang Gung Memorial Hospital (Other); Chang Gung Memorial Hospital, Chiayi (Unknown); Taoyuan General Hospital, Ministry of Health and Welfare (Unknown); Mackay Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: T3221
Record Dates: First submitted 2021-08-09; First posted 2021-09-05 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Biliary Tract Cancer (BTC)
Keywords: biliary tract cancer; Next-generation sequencing; precision medicine
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Oncopanel test
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: next-generation sequencing — Tumor tissue will be collected from advanced BTC patients for real-time next-generation sequencing analysis

SUMMARY:
Recent progress in comprehensive genomic profiling for advanced BTC has helped to clarify tumorigenesis and facilitate the coming era of precision medicine. To further elucidate the underlying molecular genomic aberrations, as well as the clinical demographics and therapeutic outcomes, it is necessary to have a national, multi-centers and population-focused research project to collect data completely. Tumor tissue will be collected from advanced BTC patients for real-time next-generation sequencing analysis in a platform of data storage and sharing. The purpose of the precision medicine project is to establish tumor molecular profiling of BTC populations in Taiwan, to facilitate patients to have corresponding potential targeted therapeutics and suitable clinical trials.

DETAILED DESCRIPTION:
Biliary tract cancer (BTC) compromises a heterogenous group of tumors with poor prognoses. Curative surgery remains the first choice for localized disease; however, most BTC patients had unresectable or metastatic disease. The gold standard therapy for these patients is chemotherapy with gemcitabine and cisplatin. There are no consensus guidelines for standard treatment in a second-line setting, although the data of the ABC-06 trial showed a slight survival benefit from oxaliplatin and 5-fluorouracil combination chemotherapy.

Recent progress in comprehensive genomic profiling for advanced BTC has helped to clarify tumorigenesis and facilitate the coming era of precision medicine. To further elucidate the underlying molecular genomic aberrations, as well as the clinical demographics and therapeutic outcomes, it is necessary to have a national, multi-centers and population-focused research project to collect data completely. Tumor tissue will be collected from advanced BTC patients for real-time next-generation sequencing analysis in a platform of data storage and sharing. The purpose of the precision medicine project is to establish tumor molecular profiling of BTC populations in Taiwan, to facilitate patients to have corresponding potential targeted therapeutics and suitable clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 20 and above.
2. Pathological reported showed adenocarcinoma or adenosquamous carcinoma for patients with BTC (include IHCC, EHCC, GBC or AVC) or hepatocholangiocarcinoma as locally advanced or metastatic status.
3. Willingness to provide the residual biopsy/operative slides.
4. Life expectancy more than 3 months.
5. Patients fully understand the protocol with the willingness to have regular follow-up.
6. Patients are ready to have 1st systemic treatment or under 1st line therapy
7. Total bilirubin ≦5 mg/dL, and ECOG≦2

Exclusion Criteria:

1. Inability to cooperate by providing a complete medical history.
2. No available tumor tissues for genetic testing.
3. Undesirable compliance.
4. Other malignancy within the past 1 years except adequately treated basal or squamous cell skin cancer or cervical cancer in situ.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ready to have 1st systemic treatment or under 1st line therapy therapy, metastatic or unresectable population s , clinical information , and therapeutic outcomes in advanced BTC
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
To enroll 400 patients who fit the criteria of this study in the enrolled period | 5 years
  To enroll 400 patients who fit the criteria of this study in the enrolled period
To perform large-scale NGS analysis for specific populations | 5 years
  To create a map containing important genetic characteristics

SECONDARY OUTCOMES:
Collect clinical data of Biliary tract cancer patients | 5 years
  Collect clinical data of Biliary tract cancer patients
To correlate the clinical characteristics, treatment and outcome of Biliary tract cancer with the genetic profile in Taiwan. | 5 years
  To correlate the clinical characteristics, treatment and outcome of Biliary tract cancer patients

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, MD, Study Chair — National Health Research Institutes, Taiwan; Ming-Huang Chen, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan; Nai-Jung Chiang, MD, PhD, Principal Investigator — National Health Research Institutes, Taiwan
Locations (13):
- Taiwan (13):
  - Chang Gung Memorial Hospital, Chiayi, Chiayi City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital,, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - MacKay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University-Shuang Ho Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Linko Chang Gung Memorial Hospital, Taoyuan District
  - Taoyuan General Hospital, Ministry of Health and Welfare, Taoyuan District

IPD SHARING:
Plan to Share IPD: No